CLINICAL TRIAL: NCT05120167
Title: Strategies for Endocervical Canal Investigation in Women With Abnormal Screening Cytology (ASC-H+) and Negative Colposcopy
Brief Title: Strategies for Endocervical Canal Investigation in Women With Abnormal Screening Cytology and Negative Colposcopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cirbia Silva Campos Teixeira (Other)
Responsible Party: Sponsor-Investigator, Cirbia Silva Campos Teixeira, Medical Doctor, Barretos Cancer Hospital
Organization: Barretos Cancer Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 49006721.5.0000.5437
Record Dates: First submitted 2021-10-17; First posted 2021-11-15 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Diagnoses Disease; Screening; HSIL of Cervix; Cervical Cancer
Keywords: Diagnostic Methods; Additional Endocervical Brushing; Endocervical canal curettage; Screening and Prevention Cervical Cancer; Precancer lesion
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Study design Clinical, randomized, controlled trial to evaluate the performance of tests for diagnosing precursor and invasive lesions in the endocervical canal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Endocervical cytology performed by liquid-based cytology (Active Comparator): Endocervical sample collected by brushing and preserved in a liquid base, and evaluated as cytology.
  Interventions: Diagnostic Test: Endocervical liquid-base cytology
- Endocervical cell block from a canal sample preserved in a buffered formalin base (Active Comparator): Endocervical sample collected by brushing and preserved in a buffered formalin base for obtaining a "cell block", and evaluated similarly as histology.
  Interventions: Diagnostic Test: Endocervical cell block
- Endocervical curettage (Active Comparator): Endocervical curettage sample preserved in buffered formalin and evaluated by histology.
  Interventions: Diagnostic Test: Endocervical curettage

INTERVENTIONS:
Diagnostic Test: Endocervical liquid-base cytology — Endocervical sample collected by brushing and preserved in a liquid-base.
  Arms: Endocervical cytology performed by liquid-based cytology
Diagnostic Test: Endocervical cell block — Endocervical sample collected by endocervical brush and preserved in a buffered formalin base for obtaining a "cell block" and evaluated as histology.
  Arms: Endocervical cell block from a canal sample preserved in a buffered formalin base
Diagnostic Test: Endocervical curettage — Endocervical sample obtained by curettage, preserved in buffered formalin, and evaluated as histology.
  Arms: Endocervical curettage

SUMMARY:
cervical cancer is the fourth most frequent cancer in women worldwide and in Brazil, it occupies the third position for the triennium 2020/2022, with a high mortality rate and maintained in the last 10 years. It is associated with persistent human papillomavirus (HPV) infection. Primary prevention can be accomplished through vaccines that prevent HPV infection of the epithelial cells of the cervix. Secondary prevention in screening for precursor lesions through periodic repeat cervical sampling in a population of asymptomatic women. Women with abnormal cytology are more likely to have pre-invasive or invasive lesions and are referred for further testing, colposcopy. Colposcopy identifies suspicious areas and guides the best site for biopsy. In the situation of negative colposcopy and abnormal cytology, suspicion for high-grade lesion (HSIL). It recommends further investigation of the endocervical canal before the possible excisional procedure and obtaining an additional canal sample by brushing or curettage. However, to date, there is no consensus and studies lack consistent results on which is the best method for further investigation of the endocervix. Objectives: To compare the performance of additional strategies in the investigation and detection of precursor or invasive lesions in the endocervical canal in women with abnormal cytology (ASC H+) and with initial colposcopy without suspicious images.

DETAILED DESCRIPTION:
Cervical cancer is a serious public health problem, with high incidence and mortality rates, especially in places with lower Human Development Index (HDI) and less access to preventive health actions and uterus has as a necessary factor a persistent infection by Human Papillomavirus (HPV), which can be detected in more than 99% of cases. There are at least 15 related to cervical cancer. These HPVs are called high-risk oncogenic HPV (HR-HPV). There is a long period of evolution from infection, its persistence resulting in the precursor lesions to the development of the invasive phase of the disease. Prevention of cervical cancer can be accomplished primarily through vaccines that prevent HPV infection of the epithelial cells of the cervix. Another form of cervical cancer prevention, called secondary prevention, is based on screening for precursor lesions through periodic repeat cervical sampling in a population of asymptomatic women. The most widely used test in the world is the conventional cytology, the so-called Papanicolaou or preventive. More recently, some countries have adopted the research of HPV DNA in samples collected in a similar way to the cytology but deposited in a liquid medium, which allows, depending on the situation, the cytological exam to be performed in the same material. Periodic screening allows for the identification of women with changes in the tests that indicate a higher risk of presenting precursor lesions and referral for treatment of lesions still in the pre-invasive phase of the disease. The Brazilian guidelines for cervical cancer screening of the Ministry of Health in 2016 recommend the periodic repetition of conventional cytological smear in women between the age group of 25 to 64 years, after initiation of sexual activity, and with a three-year interval, after two consecutive tests, with an annual interval, normal. Women diagnosed with abnormal cytology, according to country-specific scientific guidelines, following the precepts of higher risk probability for the presence of pre-invasive or invasive lesions, are referred for complementary propaedeutic with a colposcopy. Colposcopy is a visual inspection examination of the cervix with a magnifying lens, under adequate lighting, and using special reagents such as acetic acid, considered indispensable, and iodine-containing solutions such as Schiller's solution. The goal of colposcopy is to identify suspicious areas of abnormality on the surface of the cervix, guiding the best site for cervical biopsy to obtain histopathological confirmation for an initial evaluation of the extent of the lesions, information that is essential for planning the next steps. The identification of the transformation zone (TZ) by colposcopy is considered a key point in assessing the validity of colposcopic findings. It is the region of highest risk for the emergence of HPV-induced lesions and the formation of precursor lesions. The TZ needs to be visible and classified to certify the validity of the colposcopy results and to flag possible difficulties in interpreting the results and defining the best diagnostic and therapeutic approach. The current classification of the TZ is based on the visibility of the squamocolumnar junction (SCJ). When JEC is totally visible and in the ectocervix, it is classified as ZT type 1 (ZT1), and when JEC is totally visible and has both ectocervical and endocervical components, it is classified as ZT type 2 (ZT2). When the ZT has JEC not visible or partially visible in the endocervical canal, it is classified as ZT type 3 (ZT3). In situations with an indication of excisional procedure of the ZT, either for diagnosis or treatment, the type of ZT guides the realization of the excisional procedure, because, in the type 1 ZT, the excision must have a depth up to 1.0 cm (EZT1); when ZT type 2, excision with a depth between 1.5 to 2 cm (EZT2); and when ZT type 3, excision with a depth between 2 to 2.5 cm (EZT3) or classic conization. Although the general guidelines assist in the management of most cases, a frequent situation in daily practice is the difficulty in colposcopically investigating lesions of endocervical location. The most common situation is a colposcopy indicated by abnormal cytology, such as ASC-H+ (atypical squamous cells of undetermined significance, unable to exclude high-grade lesion or worse) and no abnormal colposcopic findings in the uterine cervix and vagina. In this situation of discordance between cytology and colposcopy, and the presence of ZT3. According to the Brazilian guidelines, by consensus of specialists, it is recommended to perform an additional investigation of the endocervical canal, before the possible indication of the excisional procedure type 3 (EZT 3) or the classic conization. For this initial evaluation of the endocervical canal, although studies show similar evidence of diagnostic performance between the additional brushing and curettage techniques. The first option would be to collect an additional sample from the endocervical canal by brushing for cytological evaluation, a technique that is easier to perform, less invasive, less painful, and has a lower rate of unsatisfactory sampling. The second option would be the collection through a curettage and sample fixed in buffered formalin and subsequent histopathological evaluation. But this technique is more difficult to perform, has a higher rate of unsatisfactory sampling, is more painful, and depends on the experience of the service. n this line, some countries or laboratories, can analyze additional sample by endocervical brush sample fixed in buffered formalin, still uncommon in Brazil in the following way: centrifugation of the formalized material, separation of the cells, and inclusion of the cellular aggregate in paraffin, called "cell block" and processed as it is done for histological evaluation. More recently, the emergence of new diagnostic tools, such as liquid-based cytology, the use of HPV DNA testing, p16 and Ki-67 biomarkers, are being studied in how to participate in the investigation of altered screening tests and may add information in the investigation of possible endocervical lesions. In cases of difficulties in the colposcopic assessment specified above. These new tests, in association with additional repeat cytology or endocervical canal curettage, could help in identifying women most likely to encounter high-grade cervical intraepithelial lesions or cancer, decreasing colposcopy false-positive and false-negative cytology. These additional approaches allow for a more streamlined flowchart, with less risk of iatrogenic or unnecessary excisional procedures. These additional approaches allow for a more streamlined flowchart, with less risk of iatrogenic or unnecessary excisional procedures. Optimize the resources of investigation strategies and minimize adverse effects on the woman's physical and emotional sphere during the investigation process. The 2016 Brazilian guidelines recommend excluding the vaginal lesion and performing an endocervical canal investigation before performing the excisional procedure upon discordance between high-grade cytology and a normal colposcopy.In the same vein, the American Society for Colposcopy and Cervical Pathology (ASCCP) 2019 has a guideline in this regard. It guides the preference of performing endocervical curettage in non-pregnant patients with inadequate colposcopy, at risk situation, and no lesion identified. It recommends colposcopy and endocervical sampling upon atypia of glandular cells and the performance of an excision of the ZT type 3 (EZT3), i.e., excision with a greater extension and depth of the canal and may lead to several future complications, such as increased future obstetric risk, canal stenosis, make follow-up difficult, either by colposcopy or cytology. To date, there is controversy among experts. Scientific studies do not present consistent results about which exam presents better diagnostic performance. Either additional endocervical brushing for cytology. Whether endocervical curettage or even, the use of additional biomolecular tests, before the indication of an excisional procedure. Hypothesis: 1. the performance of liquid-based cytology sample (endocervical brush sample) will be similar to that of buffered formalin-fixed cytology evaluated by means of "cell block";2. the evaluation of the "cell block" obtained from the endocervical brush sample was feasible and obtained a good accuracy. Compared to liquid-based cytology;3. The evaluation of sample obtained by endocervical curettage will be important in diagnosis for about 20% of the evaluated cases;4. The performance of HPV DNA research of liquid-based cervical cytology will be better when associated with other investigation methods: liquid-based cytology, "cell block" or endocervical curettage;5. The performance of p16 and Ki-67 biomarkers in endocervical samples will be crucial in defining the diagnosis when the other methods were insufficient. Primary Objective: To compare the performance of additional strategies in detecting precursor or invasive lesions in the endocervical canal in women with screening cytology with ASC-H or worse and with initial colposcopy without suspicious images in cervix and vagina Secondary Objective: To evaluate the performance of the following strategies in the investigation of the endocervical canal according to the final diagnosis:1. Liquid preserved endocervical brush cytology;2. "cell block" obtained from buffered formalin-fixed endocervical brush;3. The sample obtained from endocervical curettage;4. HPV DNA research performed on the liquid-based cervical cytology performed at the initial evaluation;5. Detection of p16 and Ki-67 biomarkers in the liquid-based cytology, and of p16 in the "cell block" and in the endocervical curettage.

Data Analysis Methodology: The information bank generated by Red Cap will be reviewed to assess possible inconsistencies or filling errors that will be corrected using the original information recorded in the medical records. The final digital spreadsheet will be worked on to replace the identification of the subjects with an order number. Only the researchers will know the origin of the information. This final spreadsheet without identification will be used for statistical analysis. Initially, a descriptive statistical analysis will be performed with the calculation of proportions and the respective 95% confidence intervals (95% CI) for the variables studied and their categories, according to the additional diagnostic methods and the final diagnosis. For the descriptive analysis, the chi-square and Fisher tests will be used, when appropriate, considering a p-value less than 0.05 for statistical significance. Next, a diagnostic test type analysis will be performed with the calculation of sensitivity (SENS), specificity (SPEC), negative predictive value (NPV), and positive predictive value (PPV) of each additional procedure in defining the final diagnosis. The accuracy of the various associations between the methods will be tested. The G*Power v. 3.1.9.2 software will be used to carry out these statistical procedures. Histology or 12-month follow-up, at semi-annual intervals, with negative colposcopy and cytology results will be used as the gold standard for test performance.

ELIGIBILITY:
Inclusion Criteria:

* women aged 25 years or older with altered cytology (ASC-H+) and attended the care unit and who consented to participate in the study by signing the Informed Consent Form
* Non-pregnant

Exclusion Criteria:

* colposcopy with abnormal findings;
* total hysterectomy (extirpation of the cervix);
* cervical stenosis or imperviousness near the external orifice.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with abnormal cytology of the uterine cervix in the cervical cancer screening program
Enrollment: 288 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Acuracy of endocervical cytology sample preserved in a liquid-based in the evaluation of the endocervical canal | 12 months
  calculation sensitivity (SENS), specificity (SPEC), negative predictive value (NPV) and positive predictive value (PPV) of cytology in the diagnosis of pre-invasive and invasive cervical lesion, considering histology as the gold standard or 12-month follow-up.
Acuracy of endocervical cell block sample preserved in a buffered formalin base in the evaluation of the endocervical canal | 12 months
  calculation sensitivity (SENS), specificity (SPEC), negative predictive value (NPV) and positive predictive value (PPV) of endocervical cell block in the diagnosis of pre-invasive and invasive cervical lesion, considering histology as the gold standard or 12-month follow-up.
Acuracy of endocervical curettage sample preserved in a buffered formalin base in the evaluation of the endocervical canal | 12 months
  calculation sensitivity (SENS), specificity (SPEC), negative predictive value (NPV) and positive predictive value (PPV) of endocervical curettage in the diagnosis of pre-invasive and invasive cervical lesion, considering histology as the gold standard or 12-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Cirbia SC Teixeira, MD, Principal Investigator — Hospital de Cancer de Barretos
Locations (4):
- Brazil (4):
  - Hospital de Cancer de Barretos, Campo Grande, Mato Grosso do Sul
  - Sandra Moretti Jusselino Maniçoba Palopoli, Nova Andradina, Mato Grosso do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Hospital de Cancer de Barretos, Campinas, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lei J, Ploner A, Elfstrom KM, Wang J, Roth A, Fang F, Sundstrom K, Dillner J, Sparen P. HPV Vaccination and the Risk of Invasive Cervical Cancer. N Engl J Med. 2020 Oct 1;383(14):1340-1348. doi: 10.1056/NEJMoa1917338. PMID 32997908
- [Background] Possati-Resende JC, Fregnani JH, Kerr LM, Mauad EC, Longatto-Filho A, Scapulatempo-Neto C. The Accuracy of p16/Ki-67 and HPV Test in the Detection of CIN2/3 in Women Diagnosed with ASC-US or LSIL. PLoS One. 2015 Jul 31;10(7):e0134445. doi: 10.1371/journal.pone.0134445. eCollection 2015. PMID 26230097
- [Background] Walboomers JM, Jacobs MV, Manos MM, Bosch FX, Kummer JA, Shah KV, Snijders PJ, Peto J, Meijer CJ, Munoz N. Human papillomavirus is a necessary cause of invasive cervical cancer worldwide. J Pathol. 1999 Sep;189(1):12-9. doi: 10.1002/(SICI)1096-9896(199909)189:13.0.CO;2-F. PMID 10451482
- [Background] Burd EM. Human papillomavirus and cervical cancer. Clin Microbiol Rev. 2003 Jan;16(1):1-17. doi: 10.1128/CMR.16.1.1-17.2003. PMID 12525422
- [Background] Smith JS, Lindsay L, Hoots B, Keys J, Franceschi S, Winer R, Clifford GM. Human papillomavirus type distribution in invasive cervical cancer and high-grade cervical lesions: a meta-analysis update. Int J Cancer. 2007 Aug 1;121(3):621-32. doi: 10.1002/ijc.22527. PMID 17405118
- [Background] Munoz N, Bosch FX, Castellsague X, Diaz M, de Sanjose S, Hammouda D, Shah KV, Meijer CJ. Against which human papillomavirus types shall we vaccinate and screen? The international perspective. Int J Cancer. 2004 Aug 20;111(2):278-85. doi: 10.1002/ijc.20244. PMID 15197783
- [Background] Zeferino LC, Derchain SF. Cervical cancer in the developing world. Best Pract Res Clin Obstet Gynaecol. 2006 Jun;20(3):339-54. doi: 10.1016/j.bpobgyn.2006.01.018. Epub 2006 Mar 24. PMID 16563869
- [Background] Kjaer SK, van den Brule AJ, Paull G, Svare EI, Sherman ME, Thomsen BL, Suntum M, Bock JE, Poll PA, Meijer CJ. Type specific persistence of high risk human papillomavirus (HPV) as indicator of high grade cervical squamous intraepithelial lesions in young women: population based prospective follow up study. BMJ. 2002 Sep 14;325(7364):572. doi: 10.1136/bmj.325.7364.572. PMID 12228133
- [Background] Hall MT, Simms KT, Lew JB, Smith MA, Brotherton JM, Saville M, Frazer IH, Canfell K. The projected timeframe until cervical cancer elimination in Australia: a modelling study. Lancet Public Health. 2019 Jan;4(1):e19-e27. doi: 10.1016/S2468-2667(18)30183-X. Epub 2018 Oct 2. PMID 30291040
- [Background] Derchain S, Teixeira JC, Zeferino LC. Organized, Population-based Cervical Cancer Screening Program: It Would Be a Good Time for Brazil Now. Rev Bras Ginecol Obstet. 2016 Apr;38(4):161-3. doi: 10.1055/s-0036-1582399. Epub 2016 Apr 18. No abstract available. PMID 27088706
- [Background] El-Zein M, Gotlieb W, Gilbert L, Hemmings R, Behr MA, Franco EL; STAIN-IT Study Group. Dual staining for p16/Ki-67 to detect high-grade cervical lesions: Results from the Screening Triage Ascertaining Intraepithelial Neoplasia by Immunostain Testing study. Int J Cancer. 2021 Jan 15;148(2):492-501. doi: 10.1002/ijc.33250. Epub 2020 Aug 24. PMID 32781481
- [Background] Fonseca FV, Tomasich FD, Jung JE, Maestri CA, Carvalho NS. The role of P16ink4a and P53 immunostaining in predicting recurrence of HG-CIN after conization treatment. Rev Col Bras Cir. 2016 Feb;43(1):35-41. doi: 10.1590/0100-69912016001008. English, Portuguese. PMID 27096855
- [Background] Waxman AG, Chelmow D, Darragh TM, Lawson H, Moscicki AB. Revised terminology for cervical histopathology and its implications for management of high-grade squamous intraepithelial lesions of the cervix. Obstet Gynecol. 2012 Dec;120(6):1465-71. doi: 10.1097/aog.0b013e31827001d5. PMID 23168774
- [Background] Goksedef BP, Api M, Kaya O, Gorgen H, Tarlaci A, Cetin A. Diagnostic accuracy of two endocervical sampling method: randomized controlled trial. Arch Gynecol Obstet. 2013 Jan;287(1):117-22. doi: 10.1007/s00404-012-2542-9. Epub 2012 Sep 5. PMID 22948805
- [Background] Tuon FF, Bittencourt MS, Panichi MA, Pinto AP. [Sensibility and specificity of cytology and colposcopy exams with the histological evaluation of cervical intraepithelial lesions]. Rev Assoc Med Bras (1992). 2002 Apr-Jun;48(2):140-4. doi: 10.1590/s0104-42302002000200033. Portuguese. PMID 12205531
- [Background] Undurraga M, Catarino R, Navarria I, Ibrahim Y, Puget E, Royannez Drevard I, Pache JC, Tille JC, Petignat P. User perception of endocervical sampling: A randomized comparison of endocervical evaluation with the curette vs cytobrush. PLoS One. 2017 Nov 6;12(11):e0186812. doi: 10.1371/journal.pone.0186812. eCollection 2017. PMID 29107949
- See also: Organization WH. International Agency for Reseach on Cancer. Cervix uteri Source: Globocan 2020. Internet, 2020. — http://gco.iarc.fr/today/data/factsheets/cancers/23-Cervix-uteri-fact-sheet.pdf
- See also: Brasil. Ministério da Saúde. Instituto Nacional de Câncer. Estimativa para 2020-22 do câncer do colo uterino no Brasil e diferentes regiões, 2020. — https://www.inca.gov.br/sites/ufu.sti.inca.local/files/media/document/estimativa-2020-incidencia-de-cancer-no-brasil.pdf
- See also: ABPTGIC. Associação Brasileira de Patologia do Trato Genital Inferior e Colposcopia. Novas estratégias para o rastreamento cervical baseadas no teste para hpv, 2021. — https://colposcopiasp.org.br/boletim/boletim-no-25/novas-estrategias-para-o-rastreamento-cervical-baseadas-no-teste-para-hpv/
- See also: FEBRASGO. Federação Brasileira das Associações de Ginecologia e Obstetrícia Internet. Rastreamento para câncer de colo uterino: o que há de novo?, 2020. — https://www.febrasgo.org.br/pt/noticias/item/156-rastreamento-para-cancer-de-colo-uterino-o-que-ha-de-novo
- See also: Brasil. Ministério da Saúde. Instituto Nacional de Câncer. Diretrizes para o rastreamento do Câncer do Colo do útero. Rio de Janeiro: INCA, 2016, 2016. — https://www.inca.gov.br/sites/ufu.sti.inca.local/files/media/document/diretrizesparaorastreamentodocancerdocolodoutero_2016_corrigido.pdf
- See also: ASCCP Risk-Based Management Consensus Guidelines Committee. 2019 ASCCP Risk-Based Management Consensus Guidelines for Abnormal Cervical Cancer Scre- ening Tests and Cancer Precursors. J Low Genit Tract Dis., 24:102 - 131, 2020. — https://www.asccp.org/management-guidelines
- See also: Miranda W, Miziara F, Saieg M, and Fronza H. Atualização Nomeclatura Brasileira para Laudos citopatológicos do colo uterino e Ano-Gentiais. Sociedade Brasileira de Citopatologia. 2020. — https://colposcopia.org.br/wp-content/uploads/2020/08/E-BOOK-SOCIEDADE-BRASILEIRA-DE-CITOPATOLOGIA_SBC-1-1.pdf
- See also: Organization WH. International Agency for Reseach on Cancer. Citopatologia do colo uterino - atlas digital: Sistema Bethesda de 2001. Internet, 2001. — https://screening.iarc.fr/atlascyto.php?lang=4
- See also: Brasil. Ministério da Saúde. Instituto Nacional de Câncer. Resolução CNS 466/12. — https://www.inca.gov.br/publicacoes/legislacao/resolucao-cns-466-12